CLINICAL TRIAL: NCT03848442
Title: Feasibility and Effectiveness of an Individualized 12-week 'Uptime' Participation Intervention (U-PART) in Girls and Women With Rett Syndrome
Brief Title: 'Uptime' Participation Intervention in Girls and Women With Rett Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Michelle Stahlhut, Research physiotherapist, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Center for RTT- 2017
Record Dates: First submitted 2019-02-08; First posted 2019-02-20 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Rett Syndrome
MeSH Terms: conditions — Rett Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- UPART intervention group (Experimental): A 1-group pretest-posttest design was conducted. Outcomes were evaluated on four occasions; twice during baseline separated by six weeks and immediately following a 12-week 'uptime' participation intervention and after a further 12 weeks (follow-up).
  Interventions: Other: 'Uptime' participation

INTERVENTIONS:
Other: 'Uptime' participation — The intervention are designed for each individual and are consistent with the model for participation-based interventions. The interventions are goal-oriented (meaningful and family/client-selected goals), family/client-centered (promoted self-determination and decision making), collaborative (partnership between caregivers), strength-based (built on participant and caregiver strengths) and ecological (natural environment and real-life experiences). Design of the intervention comprised three steps: 1) Preparation period (6 weeks); 2) Intervention period (12 weeks); 3) Follow-up period (12 weeks)

SUMMARY:
The aim of the study is to evaluate the feasibility and health-related effects of an individualized 12wk 'uptime' participation intervention in girls and women with Rett syndrome. Girls and women above 5 years of age with Rett syndrome and a confirmed MECP2 mutation will be included. Each individual program focuses on participation in enjoyable activities to promote 'uptime' in home, school/day center and community settings. Primary outcomes are sedentary time and daily steps. Secondary outcomes are gross motor skills, walking capacity, quality of life and participation-level goals. Outcomes are evaluated on four occasions: at baseline and after a 6-week interval, immediately following the 12-week intervention program and 12 weeks after the intervention program.

ELIGIBILITY:
Inclusion Criteria:

* Girls and women above 5 years of age with Rett syndrome and a confirmed MECP2 mutation
* Hoffer ambulation scale levels I-IV

Exclusion Criteria:

* Girls and women who have undergone orthopedic surgery in the lower extremities within the last 6 months
* Girls and women who have undergone spinal fusion within the last 12 months

Min Age: 5 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-02-07 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
ActivPAL | Assessed four times; twice at baseline; once after the 12 week intervention and once after a further 12 week follow-up
  Change in sedentary time
Stepwatch Activity Monitor | Assessed four times; twice at baseline; once after the 12 week intervention and once after a further 12 week follow-up
  Change in daily step count

SECONDARY OUTCOMES:
Rett Syndrome Gross Motor Scale | Assessed four times; twice at baseline; once after the 12 week intervention and once after a further 12 week follow-up
  Change in gross motor skills
2 minute walk test | Assessed four times; twice at baseline; once after the 12 week intervention and once after a further 12 week follow-up
  Change in walking capacity
Quality of Life Inventory - Disability, questionnaire | Assessed four times; twice at baseline; once after the 12 week intervention and once after a further 12 week follow-up
  Change in quality of life. The Quality of Life Inventory-Disability was used to assess quality of life. This 32 item-questionnaire was developed for children 5-18 years of age with ID. Responses are used to calculate an overall score and six subscale scores (social interaction, positive emotions, physical health, negative emotions, leisure/outdoors and independence), each scored on a 0-100 scale with higher scores representing better quality of life.
Goal attainment scaling | Assessed twice; at baseline and after the 12 week intervention
  Change in participation level goals. Goal attainment scaling is a validated method for evaluating achievement of individual goals. Individual goals were assessed on a five-point rating scale ranging from -2 to +2. Baseline was set at -2, the expected level after the intervention at zero and the most favorable outcome at +2. The goals were graded in relation to frequency or duration of an activity.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Rett syndrome, Department of Paediatrics and Adolescents Medicine, Copenhagen, København Ø, Denmark

IPD SHARING:
Plan to Share IPD: No